CLINICAL TRIAL: NCT01091506
Title: A Placebo-Controlled Study of Physiologic Effects of L-methylfolate in Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamlab, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: D-003
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2015-01

CONDITIONS: Schizophrenia
Keywords: L-methylfolate; Deplin; schizophrenia; folate; folic acid; homocysteine; methionine; MTHFR genotype; C677T mutation; vitamin B6; vitamin B12; psychotic symptoms; MTHFR C677T Polymorphism
MeSH Terms: conditions — Schizophrenia | interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-methylfolate (Experimental): L-methylfolate 15mg (a medical food)
  Interventions: Other: L-methylfolate
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo once a day for 12 weeks
  Arms: Placebo
Other: L-methylfolate — L-methylfolate 15mg once a day for 12 weeks
  Other Names: Deplin
  Arms: L-methylfolate

SUMMARY:
This study is a 12-week, double-blind, placebo-controlled trial of L-methylfolate 15 mg/d supplementation in schizophrenia patients with mild or greater negative symptoms. L-methylfolate, a prescription medical food, is the activated form of folate required for conversion of homocysteine to methionine and hence is the optimal form of folate for supplementation, since it eliminates the need for activation by MTHFR. The purpose of this study is to examine the change in plasma L-methylfolate concentrations following a three-month trial of L-methylfolate 15 mg/d compared to placebo.

DETAILED DESCRIPTION:
Blood levels of L-methylfolate and biological activity will be evaluated by examining changes in plasma homocysteine concentrations, serum methionine concentrations and changes in brain activation as measured by fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, any subtype
* Male of female
* Age 18-68 years
* Treated with an antipsychotic for at least 6 months at a stable dose for at least 6 weeks
* PANSS total score of at least 60, with at least 3 (moderate) on one negative symptom item or on one positive symptom item
* Simpson Angus Scale (SAS) for the EPS total score of 12 or less and
* A score of 2 (mild) or less on all items of the Calgary Depression Rating Scale (CDRS)
* Comprehension of English adequate to complete cognitive testing

Exclusion Criteria:

* Unable to provide informed consent
* CBC results consistent with megaloblastic anemia
* Serum creatinine concentration greater than 1.4
* Current use of folate supplementation > 400mcg folate
* Alcohol or other substance abuse within 3 months (nicotine allowed)
* Current use of any of the following medications: phenobarbital, phenytoin, carbamazepine, valproic acid, fosphenytoin, primidone or pyrimethamine
* Positive baseline urine toxic screen, (positive test for PCP, barbiturates, cannabinoids, amphetamines, benzodiazepines, opiates, or cocaine)
* Unstable medical illness (exclusionary lab values are listed in Appendix A)
* Unstable psychiatric illness
* Seizure disorder
* Pregnant or nursing, or planning/trying to get pregnant within the next 6 months, and
* DSM-IV diagnosis of major depressive disorder

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Examine the change in plasma L-methylfolate concentrations following a three-month trial of L-methylfolate 15 mg/d compared to placebo. | Weeks 2, 8, and 12

SECONDARY OUTCOMES:
Examine the change in brain activation in patients receiving L-methylfolate 15 mg/d versus placebo as measured by fMRI using Sternberg's Iterm Recognition Paradigm, as well as changes in cortical thickness and connectivity. | Week 12
Examine the relationship between MTHFR genotype, change in plasma homocysteine, and methionine concentration, and change in DLPC activation in subjects receiving L-methylfolate | Weeks 2, 8, and 12
Examine the change in negative symptoms (SANS total score) after three months compared to placebo | Weeks 2, 8, and 12
Examine the change in negative symptoms (SANS total score) in relation to change in plasma L-methylfolate levels | Weeks 2, 8, and 12
Examine the change in MATRICS cognitive battery composite score after three months compared to placebo | Weeks 2, 8, and 12
Examine the change in MATRICS cognitive battery composite score after three months in relation to change in plasma L-methylfolate concentration. | Weeks 2, 8, and 12
Examine the change in psychotic symptoms as measured by the PANSS total and subscale scores after three months compared to placebo | Weeks 2, 8, and 12
Examine the change in psychotic symptoms (PANSS score) in relation to change in plasma L-methylfolate concentration. | Weeks 2, 8, and 12
Examine the change in plasma homocysteine and methionine concentrations following a three-month trial of L-methylfolate 15 mg/d compared to placebo. | Weeks 2, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Roffman, MD, Principal Investigator — Massachusetts General Hospital Schizophrenia Program at Freedom Trail Clinic
Locations (1):
- Massachusetts General Hospital (MGH) Schizophrenia Program at Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Roffman JL, Petruzzi LJ, Tanner AS, Brown HE, Eryilmaz H, Ho NF, Giegold M, Silverstein NJ, Bottiglieri T, Manoach DS, Smoller JW, Henderson DC, Goff DC. Biochemical, physiological and clinical effects of l-methylfolate in schizophrenia: a randomized controlled trial. Mol Psychiatry. 2018 Feb;23(2):316-322. doi: 10.1038/mp.2017.41. Epub 2017 Mar 14. PMID 28289280